CLINICAL TRIAL: NCT04789200
Title: APhase 2 Open Label, Study to Evaluate Safety, Pharmacokinetics & Efficacy of Oral Contrast Agent, NX9 for Delineation of Bowel Anatomy at CT Imaging With/Without IV Contrast in Subjects With Cancer or GI Disease Typically Evaluated With CT
Brief Title: Phase 2 Study of NX9 for Delineation of Bowel Anatomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nextrast, Inc. (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NX9-PH2-01; 5R44DK103495 (NIH)
Record Dates: First submitted 2021-03-02; First posted 2021-03-09 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: GI Carcinoma; GI Disorders
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- NX9 oral contrast agent (Experimental): Subjects will be given a 9% w/w HBGM concentration of NX9 provided as 1.2L of liquid.
  Interventions: Drug: NX9 Oral Contrast Agent

INTERVENTIONS:
Drug: NX9 Oral Contrast Agent — Distension and marking of the bowel lumen will be compared between the 1st and 2nd scan. Ability to see IV contrast enhancement will be assessed on the 3rd scan in relationship to the 2nd scan.

SUMMARY:
This study will evaluate marking and distention of the bowel of the oral contrast agent, NX9, at CT of the abdomen and pelvis, VLDCT with no contrast will be followed by VLDCT with NX9 contrast followed by CT with NX9 and standard IV contrast. Eligible subjects will have cancer or other GI disorders for which CT is typically used to assess their disease. This is an open label study with efficacy evaluated in a masked fashion following completion of the entire study. Results of the NX9 scans will not be used for treatment decisions. PK will be evaluated in a subset of subjects at a single center.

ELIGIBILITY:
Inclusion Criteria:

1. Understands the requirements of the study and provides written informed consent prior to undergoing any study-related procedures
2. Subject is between the ages of 18 to 85 years old, inclusive
3. Has had CT of the abdomen and pelvis with IV contrast within 6 months
4. Has a concern for disease involvement of the bowel or structure adjacent to bowel (e.g. peritoneal disease, carcinomatosis, omental cake, bowel inflammation, lymphadenopathy, or fluid collection).
5. Is willing and able to comply with protocol-specified CT scanning and visits to the clinic
6. Is able to lie flat with arms above head for 15 minutes and hold breath for 15 seconds
7. Is able to drink 1.2 liters of fluid within 45 minutes
8. Has good venous access as determined by the Investigator at screening
9. Is an outpatient who is able and willing to come to the clinic for study visits

Exclusion Criteria:

1. Has any co-morbidity that the Investigator judges will interfere with their ability to complete the study or undergo a quality CT scan, e.g. high risk of aspiration
2. Has a history of or is currently suffering from a known gastrointestinal motility disorder, e.g. severe constipation / gastroparesis, achalasia, pseudo-obstruction, etc.
3. Has symptoms of a possible current bowel obstruction
4. Has a moderate to high risk of current bowel perforation
5. Subject should not schedule a GI diagnostic surgery or hospitalization for any procedure until after the study follow-up on Day 14 day. However, if at the time of study entry, the subject has pre-planned a surgery or hospitalization, it may be allowed at the discretion of the PI provided it does not take place until after the subject completes the Day 3 visit.
6. Has a contraindication (i.e. allergy) to IV or Oral CT contrast
7. If of child-bearing potential, has a confirmed pregnancy or a high probability of pregnancy at the time of screening
8. Has received an investigational therapeutic or diagnostic agent or been treated with an investigational device within the 30 days prior to enrollment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Marking and distension of the bowel lumen at CT of the abdomen | approximately 30 minutes
  Evaluated by CT imaging of the abdomen and pelvis taken in the following order: VLDCT without contrast, VLDCT with NX9 oral contrast; Readers will assess the Stomach, duodenum, jejunum, ileum, terminal ileum, proximal colon, and distal colon to record the bowel distension as the diameter of the bowel measured as mm distance from inner wall to inner wall, and the marking of bowel as the fraction of bowel length marked by NX9 contrast agent rated on a 5 point scale from 0=none, 1=0 to <25%, 2=25 to <50%, 3=50 to <75%, and 4=75 to 100% the length of the bowel.

SECONDARY OUTCOMES:
Safety: Incidence of Treatment-Emergent Adverse Events as assessed by physical exam findings and symptoms reported verbatim by subjects. | Up to 14 days
  Changes from pre-dose physical exam will be assessed by the PI and recorded as an adverse event, either related or not related to study drug. Additionally, subjects will be queried as to how they are feeling immediately following administration of study drug through 4 hours post-administration, on their Day 3 visit and during the Day 14 phone call. All symptoms will be evaluated by the PI and recorded as adverse events as appropriate. For example, if there are symptoms that are not in keeping with their pre-dose medical history.
Safety: Changes in Hematology, Chemistry and Urinalysis parameters - Screening to Post-NX9 dosing | Up to 14 days
  An abnormal laboratory result or a change from baseline will be considered an AE if it induces clinical signs or symptoms, if the abnormality is of a degree that requires active management (e.g. discontinuation of the study drug, dose modification) or when the event is requiring treatment or other therapeutic intervention (e.g. iron supplements, blood transfusion, etc.). The following parameters will be evaluated: Hematology (Hgb, RBC, WBC, Platelets, HCT), Chemistry (BUN, Creatinine, ALT, AST, GGT, LDH, AlkPhos, Total Bilirubin, Glucose, Albumin, Total Protein, Sodium, Calcium, Potassium, Phosphate, Chloride, Bicarbonate, Urate, Total Cholesterol), Urinalysis (pH, Specific gravity, Glucose, Protein, Ketones, Bilirubin, Blood, Nitrites, Leukocytes, Urobilinogen). Analysis will look for trends in clinical laboratory abnormalities.
Safety: ECGs will be used to assess clinically significant changes that may be indicative of a treatment-emergent AE. Analysis will look for overall trends in ECG changes post-dosing. | Up to 14 days
  Standard 12-lead ECGs will be taken on the Day of dosing approximately 1 hour prior to dosing and at 4 hours post-dose and on the Day 3 follow up visit. The following parameters will be recorded (Ventricular rate in bpm, PR interval, RR interval, QRS interval, QT interval, QTcF and overall reading. Any clinically significant findings and changes will be investigated by the PI and reported as AEs if appropriate.
Safety: Changes in vital signs from Screening to Post-study drug administration will be assessed for clinical significance and possibility that they are indicative of an AE. Analysis will look for overall trends in vital sign changes post-dosing. | Up to 14 days
  Standard 12-lead ECGs will be taken on the Day of dosing approximately 1 hour prior to dosing and at 4 hours post-dose and on the Day 3 follow up visit. The following parameters will be recorded (Ventricular rate in bpm, PR interval, RR interval, QRS interval, QT interval, QTcF and overall reading. Any clinically significant findings and changes will be investigated by the PI and reported as AEs if appropriate.
PK: Maximum serum concentration of NX9 following dosing will be assessed in the PK subgroup. | Up to 2 days
  Serum samples will be taken at about 2 hours pre-dose, 60 minutes post dose, 4 hours post-dose and 72 hours post dose and evaluated for Cmax.
PK: Maximum urine concentration of NX9 following dosing will be assessed in the PK subgroup. | Up to 2 days
  Urine samples will be taken at about 2 hours pre-dose, 60 minutes post dose, 4 hours post-dose and 72 hours post dose and evaluated for Cmax.
Delineation of bowel wall enhancement related to concurrent intravenous contrast at CT of the abdomen and pelvis | approximately 30 minutes
  Evaluated by CT imaging of the abdomen and pelvis taken in the following order: VLDCT without contrast, VLDCT with NX9 oral contrast; Scored on 4-point scale where 0=Cannot determine presence or absence of IV contrast enhancement of bowel wall for any of the oral contrast-filled bowel,1=IV contrast enhancement of bowel wall is clearly assessed for less than half of the oral contrast-filled bowel, 2=IV contrast enhancement of bowel wall is clearly assessed for most of the oral contrast-filled bowel, and 3=IV contrast enhancement of bowel wall is clearly assessed for all of the oral contrast-filled bowel

CONTACTS AND LOCATIONS:
Overall Officials: Michael Davis, MD, Study Director — Nextrast, Inc.
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
IPD that supports publications and presentations.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: During the review cycle for publications and presentations or post-publication when requested and approved, dependent on use of such information
Access Criteria: Written requests to be submitted to the Nextrast with plan for use of such information.